CLINICAL TRIAL: NCT04720703
Title: A Theory Driven, Rurally Tailored, Family-Based, Telehealth Intervention for Childhood Obesity: A Randomized Waitlist Controlled Trial
Brief Title: A Theory Driven, Rurally Tailored, Family-Based, Telehealth Intervention for Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Wasantha P. Jayawardene, Assistant Research Scientist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002454944
Record Dates: First submitted 2021-01-04; First posted 2021-01-22 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Childhood Obesity
Keywords: childhood obesity; telehealth; family-based
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Intervention Group will receive the Family-based Telehealth Intervention for the first three months of the study period. Once they have completed the intervention, there will be a two-week washout period. After the washout period, they will receive monthly newsletters, with similar information learned in the intervention, for three months until the end of the study period.
  Interventions: Behavioral: Family-based Telehealth Intervention
- Wait-list Control Group (Active Comparator): The Waitlist Control Group will receive monthly newsletters, with similar information learned in the intervention, for the first three months of the study period while the Intervention Group receives the intervention. Then, there will be a two-week washout period. After the washout period, they will receive the Family-based Telehealth Intervention for 3 months until the end of the study period.
  Interventions: Behavioral: Newsletters

INTERVENTIONS:
Behavioral: Newsletters — Similar to prior empirical pediatric obesity interventions (Elder et al., 2009), the active attention waitlist control group will receive monthly newsletters that focus on physical activity, healthy eating, and screen time. These newsletters will be based on standard materials from the We Can program of the National Heart, Lung, and Blood Institute (NHLBI).
  Arms: Wait-list Control Group
Behavioral: Family-based Telehealth Intervention — All communications related to the intervention will occur through weekly small group video conferencing calls via Zoom and emails or text messages. The intervention will include diverse topics proven effective in prior interventions (Davis et al., 2019; McLean et al., 2003), including reading food labels, eating out, eating at social gatherings, sticker charts, praising/rewarding healthy choices, healthy foods available at home, portion sizes, healthy/easy/low-cost cooking ideas, goal setting, monitoring screen time, exercise opportunities available in neighborhood, family exercise ideas, and healthy sleep. The research team will also send relevant video/audio clips, brochures, reminders (text messages and emails) every week.
  Arms: Intervention Group

SUMMARY:
This pilot trial aims to improve the lives of individuals in rural Indiana by addressing the leading cause of death, obesity. The purpose is to help children and their families develop healthy behaviors to decrease childhood obesity. The short-term goal of this study to develop a prototype of theory-driven, tailored, family-based, telehealth intervention that can sustainably reduce pediatric obesity rates in rural areas. The long-term goal of this study is to sustainably reduce the rates of pediatric obesity and its consequences in rural areas, via behavioral change. It is hypothesized that after participating in this intervention, children will show improvement in age-based body mass index percentile and improved behavioral indicators related to nutrition, physical activity, sleep, and sedentary behaviors. Additionally, it is hypothesized that parents will show improved attitudes and skills for managing their child's behavior and improved perceived stress and perceived quality of life. Finally, levels of attendance, participation, and technology feasibility will indicate a successful intervention.

DETAILED DESCRIPTION:
This study will utilize a purposive (non-random) sampling strategy. Children belonging to a family headed by a parent/guardian will be identified local healthcare providers practicing in any rural Indiana counties. The sampling frame will be based on the list of pediatric patients who meet eligibility criteria who currently receive services from the rural pediatric practices. Members of the research team will not have access to any medical records. Identification of the universe of eligible participants is at the sole discretion of the healthcare provider.

This study has a set of primary and secondary objectives for children and their parents/guardians, and a separate set of hypotheses for the feasibility of intervention delivery. The short-term goal is to develop a prototype for a theory-driven, tailored, family-based, telehealth intervention that can sustainably reduce pediatric obesity rates in rural areas. The long-term goal is to sustainably reduce pediatric obesity and its consequences in rural areas, solely via behavioral change.

The primary objectives for children are to improve children's behavioral indicators in terms of nutrition, physical activity, sleep, and sedentary behaviors, measured both objectively and subjectively and sustain them over time. In the end of phase-1 (at crossover point), improvement of behavioral indicators related to nutrition, physical activity, sleep, and sedentary behaviors among children who were in the intervention group will be superior to those in the control group, however, there will be no difference after phase-2 (end of study).

The secondary objective for children is to improve children's body composition, measured with the age-sex based BMI percentile. In the end of phase 1, improvement in age-sex based BMI percentile among children who were in the intervention group will be superior to those who were in the control group; however, there will be no difference after phase 2.

The primary objectives for parents/guardians are to improve caregivers' attitudes and skills, measured as constructs in the Theory of Planned Behavior (i.e., attitudes toward behavior, subjective norms, perceived behavioral control, and response efficacy), that are necessary to change their child's behaviors. In the end of phase 1, parents/guardians who were in the intervention group will show improved attitudes and skills that evidence suggests helps to change their child's behaviors, compared to those who were in the control group.

The secondary objectives for parents/guardians is to improve perceived stress and quality of life among parents/guardians. In the end of phase 1, perceived stress and perceived quality of life among parents/guardians will be better in the intervention group than the control group; however, there will be no difference after phase 2.

The tertiary objective is to assess the feasibility of the intervention at the end of the study for the intervention group only. Intervention will have the levels of attendance and participation (i.e., interaction) and technology feasibility (i.e., internet connectivity and digital literacy) required for it to be successful.

ELIGIBILITY:
Inclusion Criteria:

* 5-11 years old
* Overweight (body mass index (BMI) at or over 85th percentile, but less than 95th percentile) or Obese (BMI at or over the 95th percentile)
* living in rural Indiana
* sibling of enrolled participant - must meet all inclusion criteria with the exception of BMI

Exclusion Criteria:

* Having any of the following chronic conditions:
* developmental disabilities
* cognitive impairment
* eating disorders (e.g., anorexia nervosa, avoidant/restrictive food intake disorder, and eating disorders not elsewhere classified)
* psychiatric illnesses
* significant diagnosed medical problems (e.g., cancer) that limit physical activity, etc.
* Their only available parent parent/guardian have developmental disabilities, cognitive impairments, and psychiatric illnesses.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Intervention Attendance | 26 weeks
  Attendance to telehealth sessions will be recorded by the interventionist and calculated as a percentage for each participant. This percentage will be calculated by dividing number of sessions attended by total number of sessions.
Level of Participation | 26 weeks
  Participants are asked to complete weekly tasks (e.g. updating goal sheets) and to send researchers a picture of these updating goal sheets. Level of participation will be measured by percentage of completing these weekly tasks. This percentage will be calculated by dividing number of completed tasks by total tasks.
Parent/Guardian Satisfaction | 26 weeks
  Parent/guardian satisfaction is measured using the Telehealth Satisfaction Scale, a 10-item questionnaire with a 4-point Likert scale taken by the parent/guardian and used to evaluate their satisfaction with the technology and the intervention. Total scores range from 10-40, and higher scores indicate higher satisfaction.

SECONDARY OUTCOMES:
Change in Children's Physical Activity, Sleep Behavior, and Nutrition | Change from baseline BMI at 12 weeks
  Physical activity and sleep behaviors will be evaluated using objective measures from Fitbit activity trackers. A blinded assessor will obtain and evaluate the child's physical activity data by measuring their number of steps per day and per hour, number of active minutes, and distance in miles. All days with more than 8 hours of recorded activity will be evaluated. The child's sleep activity will be measured by their bedtime, wake up time, total sleep time, and restless minutes. The Fitbit assessor will evaluate all days with data for total sleep and nap times. The Block Kids Food Screener for assessing nutrient and food group consumption, created by NutritionQuest, will be used to measure nutrition.
Change in Children's Physical Activity, Sleep Behavior, and Nutrition | Change from 12 week BMI at 26 weeks
  Physical activity and sleep behaviors will be evaluated using objective measures from Fitbit activity trackers. A blinded assessor will obtain and evaluate the child's physical activity data by measuring their number of steps per day and per hour, number of active minutes, and distance in miles. All days with more than 8 hours of recorded activity will be evaluated. The child's sleep activity will be measured by their bedtime, wake up time, total sleep time, and restless minutes. The Fitbit assessor will evaluate all days with data for total sleep and nap times. The Block Kids Food Screener for assessing nutrient and food group consumption, created by NutritionQuest, will be used to measure nutrition .
Change in Parents' Perceived Stress and Perceived Quality of Life | Change from baseline BMI at 12 weeks
  Secondary outcomes for parents/guardians are perceived stress related to childcare and perceived quality of life. The short version Parent Stress Index (PSI) is a parent/guardian self-report with 36 items. The Perceived Quality of Life Scale (PQoL) has 19 items, each with an 11-point scale, plus a global item on happiness that is utilized for comparison purposes. These will be measured at baseline, post-intervention, and after the follow-up period.
Change in Parents' Perceived Stress and Perceived Quality of Life | Change from 12 week BMI at 26 weeks
  Secondary outcomes for parents/guardians are perceived stress related to childcare and perceived quality of life. The short version Parent Stress Index (PSI) is a parent/guardian self-report with 36 items. The Perceived Quality of Life Scale (PQoL) has 19 items, each with an 11-point scale, plus a global item on happiness that is utilized for comparison purposes. These will be measured at baseline, post-intervention, and after the follow-up period.

OTHER OUTCOMES:
Change in Children's Body Mass Index | Change from baseline BMI at 12 weeks
  The primary outcome measure for eligible child participants is change in calculated BMI z-score. Weight will be measured in pounds (to the nearest decimal) by the parents/guardians, using a digital scale. Height will be measured in inches (to the nearest decimal) by the parents/guardians, using a measuring tape. Then, these units will be converted to kilograms and meters by investigators, followed by calculation of BMI, using the formula (weight in kilograms)/ (height in meters)^2, given as kg/m^2. Subsequently, the Centers for Disease Control and Prevention's (CDC) BMI percentile chart will be used for calculating the change in BMI z-score from baseline to 3 months and from 3 months to 6 months.
Change in Children's Body Mass Index | Change from 12 week BMI at 26 weeks
  The primary outcome measure for eligible child participants is change in calculated BMI z-score. Weight will be measured in pounds (to the nearest decimal) by the parents/guardians, using a digital scale. Height will be measured in inches (to the nearest decimal) by the parents/guardians, using a measuring tape. Then, these units will be converted to kilograms and meters by investigators, followed by calculation of BMI, using the formula (weight in kilograms)/ (height in meters)^2, given as kg/m^2. Subsequently, the Centers for Disease Control and Prevention's (CDC) BMI percentile chart will be used for calculating the change in BMI z-score from baseline to 3 months and from 3 months to 6 months.
Change in Parents' Self-Reported Beliefs, Behaviors, and Attitudes | Change from baseline BMI at 12 weeks
  These primary outcome measures are derived from constructs in the Theory of Planned Behavior: behavioral beliefs, attitudes toward the behavior, normative beliefs, subjective norms, control beliefs, and perceived behavioral control. For this study, attitudes toward the given behavior, subjective norms, and perceived behavioral control will be evaluated for parents/guardians along with their behaviors that have a direct impact on the child participant's dietary, physical activity, and sleep behaviors. In addition, changes in parent/guardian response efficacy (i.e., outcome expectancy) will also be evaluated, as it is thought to influence their behaviors. A self-administered questionnaire, based on a validated instrument that has 7-point Likert-type or multiple-choice items, will be sent to parents/guardians to be used for these measures.
Change in Parents' Self-Reported Beliefs, Behaviors, and Attitudes | Change from 12 week BMI at 26 weeks
  These primary outcome measures are derived from constructs in the Theory of Planned Behavior: behavioral beliefs, attitudes toward the behavior, normative beliefs, subjective norms, control beliefs, and perceived behavioral control. For this study, attitudes toward the given behavior, subjective norms, and perceived behavioral control will be evaluated for parents/guardians along with their behaviors that have a direct impact on the child participant's dietary, physical activity, and sleep behaviors. In addition, changes in parent/guardian response efficacy (i.e., outcome expectancy) will also be evaluated, as it is thought to influence their behaviors. A self-administered questionnaire, based on a validated instrument that has 7-point Likert-type or multiple-choice items, will be sent to parents/guardians to be used for these measures.

CONTACTS AND LOCATIONS:
Overall Officials: Wasantha P Jayawardene, MD, MS, PhD, Principal Investigator — Indiana University School of Public Health-Bloomington; Mary Lynn Davis-Ajami, PhD, MBA, MS, Principal Investigator — Indiana University School of Nursing-Bloomington; Allisandra G Kummer, Study Director — Indiana University School of Public Health-Bloomington; Myat Su, Study Director — Indiana University School of Public Health Bloomington
Locations (1):
- Clinical and Translational Sciences Institute (CTSI), Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be available beginning 6 months and ending 5 years following the date of our article publication.
Access Criteria: IPD will be available to researchers who provide a methodologically sound proposal with the objective to achieve aims in the approved proposal. Proposals should be directed to wajayawa@indian.edu To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).

REFERENCES:
- [Background] Andrews KR, Silk KS, Eneli IU. Parents as health promoters: a theory of planned behavior perspective on the prevention of childhood obesity. J Health Commun. 2010 Jan;15(1):95-107. doi: 10.1080/10810730903460567. PMID 20390979
- [Background] Ayala GX, Elder JP. Qualitative methods to ensure acceptability of behavioral and social interventions to the target population. J Public Health Dent. 2011 Winter;71 Suppl 1(0 1):S69-79. doi: 10.1111/j.1752-7325.2011.00241.x. PMID 21656958
- [Background] Choi L, Liu Z, Matthews CE, Buchowski MS. Validation of accelerometer wear and nonwear time classification algorithm. Med Sci Sports Exerc. 2011 Feb;43(2):357-64. doi: 10.1249/MSS.0b013e3181ed61a3. PMID 20581716
- [Background] Davis AM, Beaver G, Dreyer Gillette M, Nelson EL, Fleming K, Swinburne Romine R, Sullivan DK, Lee R, Pettee Gabriel K, Dean K, Murray M, Faith M. iAmHealthy: Rationale, design and application of a family-based mHealth pediatric obesity intervention for rural children. Contemp Clin Trials. 2019 Mar;78:20-26. doi: 10.1016/j.cct.2019.01.001. Epub 2019 Jan 7. PMID 30630108
- [Background] Davis AM, Boles RE, James RL, Sullivan DK, Donnelly JE, Swirczynski DL, Goetz J. Health behaviors and weight status among urban and rural children. Rural Remote Health. 2008 Apr-Jun;8(2):810. Epub 2008 Apr 15. PMID 18426334
- [Background] Davis AM, James RL, Boles RE, Goetz JR, Belmont J, Malone B. The use of TeleMedicine in the treatment of paediatric obesity: feasibility and acceptability. Matern Child Nutr. 2011 Jan;7(1):71-9. doi: 10.1111/j.1740-8709.2010.00248.x. PMID 21108739
- [Background] Epstein LH, Paluch RA, Roemmich JN, Beecher MD. Family-based obesity treatment, then and now: twenty-five years of pediatric obesity treatment. Health Psychol. 2007 Jul;26(4):381-91. doi: 10.1037/0278-6133.26.4.381. PMID 17605557
- [Background] Gallagher KS, Davis AM, Malone B, Landrum Y, Black W. Treating rural pediatric obesity through telemedicine: baseline data from a randomized controlled trial. J Pediatr Psychol. 2011 Jul;36(6):687-95. doi: 10.1093/jpepsy/jsr011. Epub 2011 Mar 3. PMID 21372069
- [Background] Hunsberger M, O'Malley J, Block T, Norris JC. Relative validation of Block Kids Food Screener for dietary assessment in children and adolescents. Matern Child Nutr. 2015 Apr;11(2):260-70. doi: 10.1111/j.1740-8709.2012.00446.x. Epub 2012 Sep 24. PMID 23006452
- [Background] Marchionda DM, Slesnick N. Family therapy retention: an observation of first-session communication. J Marital Fam Ther. 2013 Jan;39(1):87-97. doi: 10.1111/j.1752-0606.2011.00279.x. Epub 2012 Feb 9. PMID 25073845
- [Background] McLean N, Griffin S, Toney K, Hardeman W. Family involvement in weight control, weight maintenance and weight-loss interventions: a systematic review of randomised trials. Int J Obes Relat Metab Disord. 2003 Sep;27(9):987-1005. doi: 10.1038/sj.ijo.0802383. PMID 12917703
- [Background] Romanzini M, Petroski EL, Ohara D, Dourado AC, Reichert FF. Calibration of ActiGraph GT3X, Actical and RT3 accelerometers in adolescents. Eur J Sport Sci. 2014;14(1):91-9. doi: 10.1080/17461391.2012.732614. Epub 2012 Oct 18. PMID 24533499
- [Background] Elder JP, Ayala GX, Slymen DJ, Arredondo EM, Campbell NR. Evaluating psychosocial and behavioral mechanisms of change in a tailored communication intervention. Health Educ Behav. 2009 Apr;36(2):366-80. doi: 10.1177/1090198107308373. Epub 2007 Dec 12. PMID 18077657
- [Background] Morgan DG, Kosteniuk J, Stewart N, O'Connell ME, Karunanayake C, Beever R. The telehealth satisfaction scale: reliability, validity, and satisfaction with telehealth in a rural memory clinic population. Telemed J E Health. 2014 Nov;20(11):997-1003. doi: 10.1089/tmj.2014.0002. Epub 2014 Oct 1. PMID 25272141